CLINICAL TRIAL: NCT03107494
Title: A Feasibility Study: A Safety Evaluation of the Gala Airway Treatment System on Patients With Chronic Bronchitis
Brief Title: Gala FIH Feasibility Study for the Treatment of Chronic Bronchitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gala Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CS002
Record Dates: First submitted 2017-03-30; First posted 2017-04-11 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Chronic Bronchitis
MeSH Terms: conditions — Bronchitis, Chronic

STUDY DESIGN:
Intervention Model Description: Treatment with Gala Airway Treatment System (RheOx)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Treatment with GATS (Experimental): Gala Airway Treatment System (GATS) / RheOx
  Interventions: Device: Gala Airway Treatment System

INTERVENTIONS:
Device: Gala Airway Treatment System — The Gala Airway Treatment system is a device-based, energy delivery system that delivers high frequency short duration energy to the airway epithelium and sub-mucosal tissue layers. The energy is delivered via a proprietary catheter through the bronchoscope. In this study, 2 treatment sessions will be delivered 1 month apart. The right lung is treated at the first treatment session and the left lung is treated at the second treatment session. A third bronchoscopy will be performed 3 months following the second treatment session where treatment is not delivered but a cryo-biopsy will be taken from the airway sites that have been treated during the two previous bronchoscopic treatment session to evaluate the effect of the treatment on the airways producing excessive mucous. Subjects will be required to submit to several tests during the study including two CT scans (lung), respiratory function tests, exercise testing.
  Other Names: GATS; RheOx

SUMMARY:
Feasibility trial (FIH) to assess the safety and clinical utility in patients with chronic bronchitis.

DETAILED DESCRIPTION:
The Gala Airway Treatment system is a device-based, energy delivery system that delivers high frequency short duration energy to the airway epithelium and sub-mucosal tissue layers. The energy is delivered via a proprietary catheter through the bronchoscope.

Two sessions of treatment will be delivered one month apart. The right lung is treated at the first treatment session and the left lung is treated at the second treatment session (approximately one month after the right side is treated). Treatment will be delivered by a respiratory physician (interventional pulmonologist) in a tertiary teaching hospital during a bronchoscopic procedure. The bronchoscopy will be delivered during general anaesthesia. It is anticipated that the bronchoscopic procedure will last less than 60 minutes in total. Treatment will be deemed to have been delivered following the successful treatment during the two bronchoscopies.

A third bronchoscopy will be performed three months following the second treatment session where treatment is not delivered but a cryo-biopsy will be taken from the airway sites that have been treated during the two previous bronchoscopic treatment session to evaluate the effect of the treatment on the airways producing excessive mucous.

Subjects will be required to submit to several tests during the study including two CT scans (lung), respiratory function tests, exercise testing.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is diagnosed with chronic bronchitis for a minimum of two years, where chronic bronchitis is defined clinically as chronic productive cough for three months in each of two successive years in a patient in whom other causes of productive cough have been excluded.
2. Subject's responses to the first two questions of the CAT must sum to at least 7 points.
3. Subject has GOLD Stage II chronic obstructive pulmonary disease (COPD) with a preprocedure post-bronchodilator FEV1 of greater than or equal to 30% and less than or equal to 80% of predicted within three months of enrollment. Subjects with a preserved function (FEV1 > 80%) are allowed if the subject has a total CAT score greater than or equal to 10 and the sum of the first two questions of the CAT score sum to at least 7 points.
4. Subject has a cigarette smoking history of at least ten packs years.
5. Subject in the opinion of the site investigator is able to adhere to and undergo three bronchoscope procedures inclusive of lung biopsies and Gala treatments and has provided a signed informed consent.

Exclusion Criteria:

1. Subject has active respiratory infection (e.g., common cold, pneumonia, MAI, tuberculosis) or COPD exacerbation within the last 6 wees prior to study treatment bronchscopy.
2. Subject is treated with > 10 mg of prednisolone or prednisone per day.
3. Subject has an implantable cardioverter defibrillator or pacemaker.
4. Subject has a history of cardiac arrhythmia within past two years.
5. Subject has abnormal cardiac rhythm at time of procedure.
6. Subject has history of proven lung cancer in last 5 years.
7. Subject has pulmonary nodule or cavity requiring follow-up or intervention unless proven benign and not actively infected (e.g., aspergilloma).
8. Subject has prior lung surgery, such as lung transplant, LVRS, lung implant/prosthesis, metal stent, valves, coils, bullectomy, segmentectomy, or lobectomy. Pneumothorax without lung resection is acceptable. Pleural procedures without surgery are acceptable.
9. Subject has Alpha-1-Antitrypsin (AAT) deficiency.
10. Subject has documented history of asthma diagnosed with onset <30 years of age, clinically significant bronchiectasis or any other significant second lung disease.
11. Subject actively smoked (including tobacco, marijuana, e-cigarettes, vaping, etc.) within the last 6 months.
12. Subject has the inability to walk over 140 meters.
13. Subject has a serious medical condition, such as: uncontrolled congestive heart failure, uncontrolled angina, myocardial infarction in the past year, renal failure, liver disease, cerebrovascular accident within the past 6 months, uncontrolled diabetes, hypertension, autoimmune disease or uncontrolled gastric reflux.
14. Subject has known sensitivity to medication required to perform bronchoscopy (such as lidocaine, atropine, and benzodiazepines).
15. Subject is pregnant, nursing, or planning to get pregnant during study duration.
16. Subject has received chemotherapy within the past 6 months or is expected to receive chemotherapy during participation in this study.
17. Subject is or has been in another clinical investigational study within 6 weeks of baseline.
18. Subject on anticoagulation for cardiovascular indications and is unable to have anticoagulants (i.e., Aspirin, Plavix, Coumadin) withheld for at least seven days prior to bronchoscopy in the opinion of the Investigator.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-01-20 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Safety: Incidence and evaluation of any serious adverse events associated with the Gala Airway Treatment System through 6 months. | 6 months
  Incidence and evaluation of any serious adverse events associated with the Gala Airway Treatment System through 6 months.

SECONDARY OUTCOMES:
Clinical Utility - Histology | 3 months following bilateral treatment
  Histopathological evidence of change in mucus producing cells within the airway.
Clinical Utility - Pulmonary Function | Through end of study (12-months post-bilateral treatment)
  Pulmonary function testing (PFT) utilizing Forced Expiratory Volume (FEV1)
Quality of Life - COPD Assessment Test (CAT) | Through end of study (12-months post-bilateral treatment)
  COPD Assessment Test (CAT) questionnaire
Quality of Life - SGRQ | Through end of study (12-months post-bilateral treatment)
  Patient filled respiratory questionnaire: St. George Respiratory Questionnaire (SGRQ)
Acute Exacerbations | From 48 hours post procedure through end of study (12 months post-bilateral treatment)
  Detection of acute exacerbations (measured by clinical examination of a suitably qualified physician)
Non-Acute Exacerbations | From 48 hours post procedure through end of study (12 months post-bilateral treatment)
  Detection of non-acute exacerbations (measured by clinical examination of a suitably qualified physician)
Six Minute Walk Test (6MWT) | 6 months post-bilateral treatment
  Change in 6MWT at 6 months compared to baseline

OTHER OUTCOMES:
Cough and Sputum Assessment Questionnaire (CASA-Q) | Through end of study (12-months post-bilateral treatment)
  Patient reported outcome respiratory questionnaire: Cough and Sputum Assessment

CONTACTS AND LOCATIONS:
Overall Officials: William Krimsky, MD, Study Director — Gala Therapeutics, Inc.
Locations (2):
- Otto Wagner Spital, Vienna, Austria
- Clinica Alemana, Santiago, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Krimsky WS, Mammarappallil JG, Kim V, Bannan B, Charbonnier JP, Hatton BA, Sciurba FC. Airway Mucus Plugging in Chronic Bronchitis and the Impact of Bronchial Rheoplasty. Chest. 2026 Jan;169(1):73-83. doi: 10.1016/j.chest.2025.06.022. Epub 2025 Jun 24. PMID 40571054
- [Derived] Krimsky WS, VanderLaan PA, Iding JS, Hunter DW, Hatton BA, Bannan B, Kim V. A quantitative method for assessing treatment-related changes within the airway mucosa in patients with chronic bronchitis. Respir Med. 2025 Jan;236:107889. doi: 10.1016/j.rmed.2024.107889. Epub 2024 Nov 28. PMID 39615802
- [Derived] Valipour A, Fernandez-Bussy S, Ing AJ, Steinfort DP, Snell GI, Williamson JP, Saghaie T, Irving LB, Dabscheck EJ, Krimsky WS, Waldstreicher J. Bronchial Rheoplasty for Treatment of Chronic Bronchitis. Twelve-Month Results from a Multicenter Clinical Trial. Am J Respir Crit Care Med. 2020 Sep 1;202(5):681-689. doi: 10.1164/rccm.201908-1546OC. PMID 32407638